CLINICAL TRIAL: NCT00006708
Title: A Randomized Phase III Trial of ICE Chemotherapy With or Without Rituximab for the Treatment of Relapsed or Refractory CD20 Expressing Aggressive B-Cell Non-Hodgkin's Lymphomas in Patients Not Suitable for High Dose Therapy and PBSCT
Brief Title: S0019 Combination Chemotherapy With or Without Rituximab in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068320; S0019 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2000-12-06; First posted 2004-03-17 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma | interventions — Filgrastim; Rituximab; Carboplatin; Etoposide; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICE Chemotherapy (Active Comparator): Etoposide 100 mg/m2 IV Days 1-3 Carboplatin AUC=5 IV Day 2 Ifosfamide 5 g/m2 IV Day 2 Mesna 5 g/m2 IV Day 2 Filgrastim 5ug/kg/day SQ Days 5-12 Q 21 days x 3 cycles
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: etoposide; Drug: ifosfamide
- Rituximab-ICE Chemotherapy (Experimental): Etoposide 100 mg/m2 IV Days 2-4 Carboplatin AUC=5 IV Day 3 Ifosfamide 5 g/m2 IV Day 3 Mesna 5 g/m2 IV Day 3 Filgrastim 5ug/kg/day SQ Days 6-13 Q 21 days x 3 cycles Rituximab 375 mg/m2 IV Days 1 and 8 Cycle 1 Rituximab 375 mg/m2 IV Day 1 Cycles 2-3
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: carboplatin; Drug: etoposide; Drug: ifosfamide

INTERVENTIONS:
Biological: filgrastim — 5 μg/kg/day subcutaneous injection on Days 5-12 every 21 days for 3 cycles.
Biological: rituximab
  Arms: Rituximab-ICE Chemotherapy
Drug: carboplatin
Drug: etoposide
Drug: ifosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known whether combination chemotherapy is more effective with or without rituximab for non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without rituximab in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the progression-free and overall survival of patients with relapsed or refractory, CD20 expressing, aggressive, B-cell non-Hodgkin's lymphoma treated with ifosfamide, carboplatin, and etoposide with or without rituximab. II. Compare the unconfirmed response rate of patients treated with these regimens. III. Determine the toxicity of ifosfamide, carboplatin, and etoposide with rituximab in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to histology (large B-cell vs other) and risk group (low/low-intermediate vs high-intermediate/high). Patients are randomized to one of two treatment arms. Arm I: Patients receive etoposide IV over 1 hour on days 1-3, carboplatin IV over 1 hour on day 2, ifosfamide IV continuously for 24 hours on day 2, and filgrastim (G-CSF) subcutaneously (SC) on days 5-12. Treatment continues every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Arm II: Patients receive rituximab IV on day 1, etoposide IV over 1 hour on days 2-4, carboplatin IV over 1 hour on day 3, ifosfamide IV continuously for 24 hours on day 3, and G-CSF SC on days 6-13. Patients also receive rituximab IV on day 8 of course 1. Treatment continues every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 376 patients (188 per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven aggressive B-cell non-Hodgkin's lymphoma that has failed prior combination chemotherapy with an anthracycline-containing regimen Eligible histologies: Diffuse large cell Small non-cleaved cell/Burkitt's lymphoma No lymphoblastic or mantle cell lymphoma First relapse or primary refractory disease Ineligible for or refused treatment with salvage chemotherapy followed by high-dose therapy and autologous stem cell rescue Documented CD20 antigen expression Measurable disease No clinical evidence of CNS involvement by lymphoma

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Other: HIV negative Not pregnant or nursing Fertile patients must use effective contraception No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No prior rituximab Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: Recovered from toxic effects of all prior therapy No other concurrent therapy unless disease progression occurs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2000-10; Primary Completion 2002-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G. Maloney, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (85):
- United States (85):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington